CLINICAL TRIAL: NCT02200120
Title: Evaluation of Catheter Placement for Renal Replacement Therapy in Patients With Acute Kidney Injury- Assessment of Dialysis Adequacy and Infection Rates
Brief Title: Evaluation of Catheter Placement for Renal Replacement Therapy in Patients With Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Sushrut S Waikar, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 99904021982
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to examine the placement, timing, associated complications, efficacy of temporary and tunneled catheters for renal replacement therapy in patient with acute kidney injury.

DETAILED DESCRIPTION:
The purpose of this study is to examine the placement, timing, associated complications, efficacy of temporary and tunneled catheters for renal replacement therapy in patient with acute kidney injury. In particular, we will be assessing renal replacement adequacy for patients on dialysis and continuous veno-venous hemofiltration by monitoring urea reduction ratios, venous and arterial pressures. We will also be monitoring infection rates. We will compare these outcomes in patients receiving tunneled catheters and patients receiving temporary catheters.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the hospital with acute kidney injury requiring renal replacement therapy

Exclusion Criteria:

* End stage renal disease
* Chronic kidney disease 5 progression to end stage renal disease
* Outside hospital catheter placement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the hospital with acute kidney injury requiring renal replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Dialysis adequacy | up to 7d after starting renal replacement therapy
  Adequacy will be measured using urea reduction ratio for patients on intermittent hemodialysis. For continuous renal replacement therapy, we will record the maximum blood flow rate achievable. These measurements/recordings will be made on average within 1-3 days of starting therapy.

SECONDARY OUTCOMES:
blood stream infection rates | within 30d of catheter placement
  Patients will be followed throughout their hospitalization, which can range from a few days to several weeks. Bloodstream infections within 30d of catheter placement will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sushrut Waikar, MD, MHS, Principal Investigator — Brigham and Women's Hospital; Mallika L Mendu, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States